CLINICAL TRIAL: NCT05778955
Title: The Significance of Dynamic Monitoring of ctDNA in Pediatric Soft Tissue Sarcoma
Brief Title: Study on Dynamic CtDNA Analysis in Pediatric Soft Tissue Sarcoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Nanjing Geneseeq Technology Inc. (Industry)
Responsible Party: Principal Investigator, Yizhuo Zhang, Director of Pediatric Oncology, Sun Yat-sen University
Other Study IDs: ctDNA-P-STS01
Record Dates: First submitted 2023-02-15; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Pediatric Soft Tissue Sarcoma
Keywords: Pediatric Soft Tissue Sarcoma; ctDNA; NGS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: detection and monitoring of cirulating tumor DNA — detection and monitoring of cirulating tumor DNA in pediatric soft tissue sarcoma

SUMMARY:
Pediatric soft tissue sarcoma is made up of different subtypes, some of which have distinct genetic alterations. Fusion variants were found in about 43% of bone and soft tissue sarcoma samples. Ewing sarcoma is characterized by recurrent chromosome translocation, with up to 95% of cases showing EWS-ETS translocation. The genetic features of the tumor can change as it spreads or shrinks, and can also be influenced by treatment.

To better understand treatment response and predict relapse early, our study collects liquid samples such as blood, bone marrow, or cerebrospinal fluid at various points during treatment. We then use next-generation sequencing to dynamically monitor the unique genetic profile of the tumor. Additionally, our research may identify new genetic targets and suggest potential treatment options.

ELIGIBILITY:
Inclusion Criteria:

* (1) pediatric patients with soft tissue sarcoma confirmed by pathology(including but not limited to rhabdomyosarcoma, Ewing sarcoma, BCOR rearrangement undifferentiated sarcoma, CIC rearrangement undifferentiated sarcoma, Epithelioid sarcoma and synovial sarcoma.
* (2)younger than 18 years old.
* (3)ECOG status: PS score0-2.
* (4)measurable lesions on CT/MRI according to RECIST 1.1 criteria : long diameter≥10mm; the longest diameter on ≥ one lymphnode ≥1.5 cm.
* (5)sufficient clinical and pathological information.
* (6)candidates can receive evaluation on time and provide samples during the trials.
* (7)candidates should be informed and provide informed consents.

Exclusion Criteria:

* Sufficient samples at baseline point can not be obtained including pre-operation plasma, tissues, bone marrow aspirate and cerebrospinal fluid.
* Plasma samples can not be obtained during monitoring.
* Ineligible candidates at the discretion of researchers.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Asian population predominates
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate to detected tumor progression by ctDNA before radiographic tumor progression | Oct,2022-Dec 2023,recruting patients; Jan 2024-Mar 2024,analyzing the genetic features in samples;Jan 2023-May 2024,follow up patients
  1. Progression-Free Survival PFS is defined as the time from randomization to progression or death.
  2. The definition of ctDNA positive samples : at least one of somatic alterations detected by 475-gene panel.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided